CLINICAL TRIAL: NCT05170204
Title: A Phase I-III, Multicenter Study Evaluating the Efficacy and Safety of Multiple Therapies in Cohorts of Patients Selected According to Biomarker Status, With Locally Advanced, Unresectable, Stage III Non-Small Cell Lung Cancer
Brief Title: A Study Evaluating the Efficacy and Safety of Multiple Therapies in Cohorts of Participants With Locally Advanced, Unresectable, Stage III Non-Small Cell Lung Cancer (NSCLC)
Acronym: HORIZON 1
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO42777; 2023-503920-14-00 (EU CTIS Number)
Record Dates: First submitted 2021-12-22; First posted 2021-12-27 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — alectinib; entrectinib; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A1: ALK-Positive (alectinib arm) (Experimental): Participants will receive alectinib 600 mg orally twice daily until completion of treatment period (3 years), or until disease progression, unacceptable toxicity, patient or physician decision to discontinue, or death, whichever occurs first
  Interventions: Drug: Alectinib
- Cohort A1: ALK-positive (durvalumab arm) (Active Comparator): Participants will receive 1500 mg of intravenous (IV) durvalumab every 4 weeks until completion of treatment period (1 year) or until disease progression, unacceptable toxicity, patient or physician decision to discontinue, or death, whichever occurs first
  Interventions: Drug: Durvalumab
- Cohort A2: ROS 1-positive (entrectinib arm) (Experimental): Participants will receive entrectinib 600 mg orally once daily until completion of treatment period (3 years), or until disease progression, unacceptable toxicity, patient or physician decision to discontinue, or death, whichever occurs first.
  Cohort A2 has been closed to enrollment.
  Interventions: Drug: Entrectinib
- Cohort A2: ROS 1-positive (durvalumab arm) (Active Comparator): Participants will receive 1500 mg of IV durvalumab every 4 weeks until completion of treatment period (1 year) or until disease progression, unacceptable toxicity, patient or physician decision to discontinue, or death, whichever occurs first
  Cohort A2 has been closed to enrollment.
  Interventions: Drug: Durvalumab

INTERVENTIONS:
Drug: Alectinib — Participants will receive oral alectinib twice daily with food.
  Arms: Cohort A1: ALK-Positive (alectinib arm)
Drug: Entrectinib — Participants will receive oral entrectinib once daily, with or without food.
  Arms: Cohort A2: ROS 1-positive (entrectinib arm)
Drug: Durvalumab — Participants will receive IV durvalumab every 4 weeks.
  Arms: Cohort A1: ALK-positive (durvalumab arm); Cohort A2: ROS 1-positive (durvalumab arm)

SUMMARY:
This study will evaluate the efficacy and safety of multiple therapies in participants with locally advanced, unresectable, Stage III NSCLC with eligible biomarker status as determined by Version 8 of the American Joint Committee on Cancer/Union for International Cancer Control NSCLC staging system.

ELIGIBILITY:
Inclusion Criteria (All Cohorts):

* Body weight >/= 30 kg at screening
* Willingness and ability to use the electronic device(s) or application(s) for the electronic patient-reported outcome (PRO)
* Whole-body positron emission tomography/computed tomography scan (PET/CT) (from the base of skull to mid-thighs) for the purposes of staging, performed prior and within 42 days for Cohort A2 (ROS1 positive) and 50 days for Cohort A1 (ALK positive) of the first dose of cCRT or sCRT
* Histologically or cytologically documented locally advanced, unresectable Stage III NSCLC of either squamous or non-squamous histology
* Prior receipt of at least two prior cycles of platinum-based chemotherapy given concurrently with radiotherapy (cCRT); or at least two prior cycles of platinum-based chemotherapy given prior to radiotherapy (sCRT)
* The RT component in the cCRT or sCRT must have been at a total dose of radiation of 60 (+/-10%) Gy (54 Gy to 66 Gy) administered by intensity-modulated radiotherapy (preferred) or three dimension (3D)-conforming technique
* No disease progression during or following platinum-based cCRT or sCRT
* Life expectancy >/= 12 weeks
* Confirmed availability of a representative formalin-fixed, paraffin-embedded (FFPE) tumor specimen
* Tumor PD-L1 status (TC score < 1% vs. >/= 1% vs. unknown) as determined using the VENTANA PD-L1 IHC SP263 assay (preferred) or the Dako PD-L1 IHC 22C3 pharmDx assay
* Eastern Cooperative Oncology Group Performance Status of 0, 1, or 2
* Adequate hematologic and end-organ function
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception, and agreement to refrain from donating eggs, as defined by the protocol
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods, and agreement to refrain from donating sperm, as defined by the protocol

Inclusion criteria specific to Cohort A1:

* Documented ALK fusion positivity by an eligible result from: centralized multiplex molecular testing of tumor tissue at the Sponsor's designated central laboratory under Study BX43361 or prior tissue-based testing performed in an accredited or certified laboratory

Inclusion criteria specific to Cohort A2:

* Documented ROS1 fusion positivity by an eligible result from: centralized multiplex molecular testing of tumor tissue at the Sponsor's designated central laboratory under Study BX43361 or available results from a Sponsor pre-approved local, appropriately validated ROS1 fusion test on tumor tissue performed in a Clinical Laboratory Improvement Amendments certified or equivalent laboratory
* Ability to swallow entrectinib intact, without chewing, crushing, or opening the capsules

Exclusion Criteria (All Cohorts):

* Any history of previous NSCLC and/or any history of prior treatment for NSCLC (patients must be newly diagnosed with unresectable Stage III disease)
* Any evidence of Stage IV disease, including, but not limited to, the following: pleural effusion, pericardial effusion, brain metastases, history of intracranial hemorrhage or spinal cord hemorrhage, bone metastases, distant metastases
* If a pleural effusion is present, the following criteria must be met to exclude malignant involvement (T4 disease): when pleural fluid is visible on both the CT scan and chest X-ray, a pleuracentesis is required to confirm that the pleural fluid is cytologically negative; participants with exudative pleural effusions are excluded regardless of cytology; participants with effusions that are minimal (i.e., not visible on chest X-ray) that are too small to safely tap are eligible
* NSCLC known to have a known or likely oncogenic-driver mutation in the EGFR gene, as identified by site local testing or Sponsor central testing
* Liver disease, characterized by any of the following: impaired excretory function (e.g., hyperbilirubinemia), synthetic function, or other conditions of decompensated liver disease, such as coagulopathy, hepatic encephalopathy, hypoalbuminemia, ascites, and bleeding from esophageal varices or active viral or active autoimmune, alcoholic, or other types of acute hepatitis
* Positive hepatitis B surface antigen (HBsAg) test at screening
* Participants known to be positive for hepatitis C virus (HCV) antibody (Ab) are excluded with the following exception: participants who are HCV Ab positive but HCV RNA negative due to prior treatment or natural resolution are eligible
* HIV infection: participants are excluded if not well-controlled as defined by the protocol
* Known active tuberculosis
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on the screening chest CT scan
* Grade >/= 2 pneumonitis from prior cCRT or sCRT
* Any Grade > 2 unresolved toxicity from prior cCRT or sCRT
* Any gastrointestinal (GI) disorder that may affect absorption of oral medications, such as malabsorption syndrome or status post-major bowel resection
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications
* Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis, with the following exceptions: participants with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study; participants with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study
* History of malignancy other than NSCLC within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death (e.g., 5-year OS rate > 90%), such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal breast carcinoma in situ, or Stage I uterine cancer
* Any concurrent chemotherapy, immunotherapy, biologic, or hormonal therapy for cancer
* Major surgical procedure, within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study
* Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin-2) within 4 weeks or 5 drug-elimination half-lives (whichever is longer) prior to initiation of study treatment
* Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during study treatment or within 5 months after the final dose of study treatment
* Treatment with investigational therapy within 28 days prior to initiation of study treatment
* Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor-alpha agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with exceptions defined by the protocol
* Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-cytotoxic T lymphocyte-associated protein 4, anti-TIGIT, anti-PD-1, and anti-PD-L1 therapeutic antibodies
* Prior allogeneic stem cell or solid organ transplantation
* Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or the follow-up period of an interventional study
* Any condition that, in the opinion of the investigator, would interfere with the evaluation of the study drug or interpretation of patient safety or study results
* Any prior Grade >/= 3 immune-mediated adverse event or any unresolved Grade > 1 immune-mediated adverse event while receiving any previous immunotherapy agent other than immune checkpoint blockade agents

Exclusion criteria specific to Cohort A1:

* Presence of clinically symptomatic interstitial lung disease or interstitial pneumonitis, including radiation pneumonitis (i.e., affecting activities of daily living or requiring therapeutic intervention)
* NSCLC known to have one or more of the following ALK point mutations, as identified by site local testing or Sponsor central testing: I1171X (where X is any other amino acid), V1180L, G1202R
* Symptomatic bradycardia
* Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina; participants with known coronary artery disease, congestive heart failure not meeting the above criteria, or left ventricular ejection fraction < 50% must be on a stable medical regimen that is optimized in the opinion of the treating physician, in consultation with a cardiologist if appropriate
* Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
* Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment
* Prior treatment with ALK inhibitors
* History of hypersensitivity to alectinib, durvalumab, or any of their excipients
* Inability to swallow oral study drug
* Known hereditary problems of galactose intolerance, a congenital lactase deficiency, or glucose-galactose malabsorption
* Pregnancy or breastfeeding, or intending to become pregnant during the study treatment or within 90 days after the final dose of alectinib or durvalumab

Exclusion criteria specific to Cohort A2:

* Symptomatic bradycardia
* Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina; participants with known coronary artery disease, congestive heart failure not meeting the above criteria, or left ventricular ejection fraction < 50% must be on a stable medical regimen that is optimized in the opinion of the treating physician, in consultation with a cardiologist if appropriate
* Left ventricular ejection fraction less than or equal to 50% observed during the screening for the study
* History of prolonged QTc interval (e.g., repeated demonstration of a QTc interval > 450 ms from ECGs performed at least 24 hours apart)
* History of additional risk factors for torsade de pointes (e.g., family history of long QT syndrome)
* Familial or personal history of congenital bone disorders or bone metabolism alterations
* Incomplete recovery from any surgery prior to the start of study treatment that would interfere with the determination of safety or efficacy of the treatment
* Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
* Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment
* Prior treatment with ROS1 inhibitors
* History of hypersensitivity to entrectinib, durvalumab, and their excipients
* Grade >/= 3 toxicities due to any prior therapy (e.g., RT) (excluding alopecia) that have not shown improvement or are not stable and are considered to interfere with current study drug
* Known hereditary problems of galactose intolerance, total lactase deficiency or glucose-galactose malabsorption
* Grade >/= 2 peripheral neuropathy
* Pregnancy or intention of becoming pregnant during study treatment, within 35 days after the final dose of entrectinib, or within 90 days after the final dose of durvalumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2032-08-21 (Estimated); Study Completion 2033-09-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From randomization to the first documented disease progression as determined by blinded independent central review (BICR) per Response Evaluation Criterial in Solid Tumors (RECIST) v1.1, or death from any cause, whichever occurs first (up to 3 years)

SECONDARY OUTCOMES:
Time to central nervous system (CNS) progression | From randomization to the first occurrence of disease progression in the CNS as determined by BICR per RECIST v1.1 (up to 3 years)
Distant metastasis-free survival (DMFS) | From randomization to the first occurrence of distant metastasis or death (whichever occurs first) as determined by BICR per RECIST v1.1 (up to 3 years)
Objective response rate (ORR), defined as the percentage of participants with measurable disease who attain a complete response (CR) or partial response (PR) as determined by the investigator per RECIST v1.1 | Up to 3 years
PFS | From randomization to the first documented disease progression as determined by the investigator per RECIST v1.1, or death from any cause, whichever occurs first (up to 3 years)
Duration of response (DOR) | From the first documented CR or PR to the first documented disease progression or death (whichever occurs first) as determined by the investigator per RECIST v1.1 (up to 3 years)
ORR, defined as the percentage of participants with measurable disease who attain a CR or PR as determined by BICR per RECIST v1.1 | Up to 3 years
DOR | From the first documented CR or PR to the first documented disease progression or death (whichever occurs first) as determined by BICR per RECIST v1.1 (up to 3 years)
Overall survival (OS) | From randomization to death from any cause (up to 5 years)
Time to CNS progression | From randomization to the first occurrence of disease progression in the CNS as determined by the investigator per RECIST v1.1 (up to 3 years)
Time-to-confirmed deterioration (TTCD) | From randomization to the first deterioration of >/= 10 points that is either maintained for two consecutive assessments or followed by death from any cause within 3 weeks (up to 3 years)
Proportion of participants who have maintained or improved baseline health as measured by the European Organisation for the Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ)-C30 physical functioning and role functioning scales | 5, 11, and 17 months
Proportion of participants who have maintained or improved from their baseline health in cough, chest pain, and dyspnea symptoms as measured using the EORTC QLQ-LC13 | 5, 11, and 17 months
Percentage of participants with adverse events (AEs) | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (45):
- United States (2):
  - Northwest Cancer Specialists, P.C., Tigard, Oregon
  - Hillman Cancer Center, Pittsburgh, Pennsylvania
- Australia (2):
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - One Clinical Research, Nedlands, Western Australia
- UZ Gent, Ghent, Belgium
- Brazil (2):
  - Hospital de Cancer de Barretos, Barretos, São Paulo
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
- RedSalud Vitacura, Santiago, Chile
- China (4):
  - Hunan Cancer Hospital, Changsha
  - Xinqiao Hospital of Third Military Medical University, Chongqing
  - Shandong Cancer Hospital, Jinan
  - Shanghai Pulmonary Hospital, Shanghai
- Colombia (2):
  - Fundación CTIC - Centro de Tratamiento e Investigación sobre Cáncer Luis Carlos Sarmiento Angulo, Bogota, D.C.
  - Hospital Universitario San Ignacio, Bogotá
- France (3):
  - Centre Francois Baclesse, Caen
  - Centre Leon Berard, Lyon
  - Hopital Nord, Marseille
- Helios Klinikum Emil von Behring GmbH, Berlin, Germany
- Italy (2):
  - IRST Istituto Scientifico Romagnolo Per Lo Studio E Cura Dei Tumori, Sede Meldola, Meldola, Emilia-Romagna
  - Asst Grande Ospedale Metropolitano Niguarda, Milan, Lombardy
- Japan (8):
  - NHO Kyushu Cancer Center, Fukuoka
  - Kurume University Hospital, Fukuoka
  - Kobe City Medical Center General Hospital, Hyōgo
  - Kagoshima University Hospital, Kagoshima
  - Kumamoto University Hospital, Kumamoto
  - Kindai University Hospital, Ōsaka-sayama
  - Juntendo University Hospital, Tokyo
  - The Cancer Institute Hospital of JFCR, Tokyo
- Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara, Jalisco, Mexico
- Dolno?l?skie Centrum Chorób P?uc we Wroc?awiu, Wroc?aw, Poland
- National Cancer Centre, Singapore, Singapore
- South Korea (6):
  - Kyungpook National University Chilgok Hospital, Daegu
  - Pusan National University Yangsan Hospital, Gyeongsangnam-do
  - Chonnam National University Hwasun Hospital, Jeollanam-do
  - Seoul National University Bundang Hospital, Seongnam-si
  - Asan Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Karolinska Universitetssjukhuset, Solna, Stockholm
- Taichung Veterans General Hospital, Taichung, Taiwan
- Thailand (4):
  - Rajavithi Hospital, Bangkok
  - Faculty of Med. Siriraj Hosp., Bangkok
  - Oncology Unit, Faculty of Medicine, Vajira Hospital, Dusit
  - Songklanagarind Hospital, Songkhla
- Christie Hospital Nhs Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing